CLINICAL TRIAL: NCT01469884
Title: A Prospective, Single-center, Open-label, Pilot Study to Investigate the Effect of Switching to Certican® in Viremia of Hepatitis C Virus in Adult Renal Allograft Recipients.
Brief Title: Effect of Switching to Certican® in Viremia of Hepatitis C Virus in Adult Renal Allograft Recipients
Acronym: CONCERVIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Valter Duro Garcia, PHYSICIAN NEPHROLOGY, Irmandade Santa Casa de Misericórdia de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CRAD001; CRAD001ABR20T (Other: NOVARTIS)
Record Dates: First submitted 2011-11-01; First posted 2011-11-10 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Renal Allograft; Hepatitis C
Keywords: Renal allograft recipients; Hepatitis C virus (HCV); Certican; Calcineurin inhibitor(tacrolimus or cyclosporin)
MeSH Terms: conditions — Hepatitis C | interventions — Everolimus; Cyclosporine; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Certican® (Experimental): Arm1(conversion):Certican®+mycophenolate+prednisone
  Interventions: Drug: Everolimus
- Tacrolimus or Cyclosporine (Active Comparator): Arm2(maintained):Tacrolimus or Cyclosporine+mycophenolate+prednisone
  Interventions: Drug: Cyclosporine; Drug: Tacrolimus

INTERVENTIONS:
Drug: Everolimus — The conversion will be performed abruptly for all patients. Calcineurin inhibitor will be discontinued one day before the day of conversion (Day 1). Everolimus will be introduced on day 1 at dose of 3 mg/d (1,5mg bid), and then everolimus trough levels will be adjusted to achieve 6-10 ng/ml.
  Arms: Certican®
Drug: Cyclosporine — Trough level should be between 100 and 200ng/ml.
  Arms: Tacrolimus or Cyclosporine
Drug: Tacrolimus — Trough level should be between 5 and 10ng/ml.
  Arms: Tacrolimus or Cyclosporine

SUMMARY:
Compare the viral load of hepatitis c virus in patients converted to certican versus patients who are maintained on calcineurin inhibitor.

DETAILED DESCRIPTION:
The infection by hepatitis C virus (HCV) is the leading cause of chronic liver disease in renal transplant recipients.

The prevalence of pretransplantation anti-HCV is 11% to 49%. The impact of HCV infection on patient survival after renal transplant remains controversial. Some studies also showed that patients undergoing renal transplantation anti-HCV positive are associated with a reduction in graft and patient survival.Chronic infection of HCV is associated with an increased number of infections.

In HCV positive renal transplant patients have been shown that there is an increase from four to seven times in HCV viremia after transplantation compared to pretransplant.

To prevent viral replication, immunosuppression must be adapted, involving a balance between control of viral replication and rejection.

Biochemically, the NS5A protein has been linked to increased replication of the hepatitis C virus through p70S6K phosphopeptides. Sirolimus as inhibitor of pathway mTOR/p70S6K reduced in vivo phosphorylation of NS5A phosphopeptides and thus viral replication. Moreover, the mTOR protein has been proven in vitron to have a protective role against apoptosis in HCV infected cells (WAGNER et al., 2010).

Wagner et al. (2010) showed a beneficial effect of sirolimus on viral recurrence monitored by transaminases and viral load as well as by histological data. They also reported the improved survival after liver transplantation due to hepatitis C for patients receiving sirolimus rather than calcineurin inhibitor-based regimens.

In the literature there have already been reported good virological control of HCV among liver transplant recipients after conversion to SRL and the reduction of hepatitis C virus recurrence (GALLEGO et al., 2009; BENEDETTOET al., 2010).

Everolimus has shown a potent inhibitor of mTOR and has been widely used as an immunosuppressive agent in kidney transplant, but no reported effects on HCV progression was found in the literature.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 years at the time of screening;
* Subjects between the first and tenth year after renal transplantation;
* Subjects with positive serology for hepatitis C;
* Subjects receiving calcineurin inhibitor (tacrolimus or cyclosporine) plus mycophenolate sodium or mofetil plus prednisone since the first month post-transplant;
* Subjects with no acute rejection episode in the last 3 month;
* Women of childbearing potential (CBP) with a negative pregnancy test at screening (urine or serum;
* Women of CBP and men with sexual partners of CBP must agree to use a medically acceptable method of contraception throughout the study. The investigator will determine which contraceptive method more effective and appropriate for each study subject. Acceptable methods of contraception include oral contraceptives, barrier methods (eg, diaphragm or condom with spermicide) and intrauterine devices.

Exclusion criteria:

* Subjects who, in the opinion of the investigator, are not able to complete the study;
* Recipients of multiple organ transplant (i.e., prior or concurrent transplantation of a non-renal allograft;
* Subjects with a calculated GFR < 30ml/min (abbreviated MDRD formula;
* Subjects with Urinary protein/creatinine > 0.5;
* Renal biopsy with score ≥ Banff grade II interstitial fibrosis and tubular atrophy (Banff 2007;
* Subjects with a history of biopsy-proven acute rejection within 12 weeks of enrollment;
* Known or suspected hypersensitivity to inhibitor of mTOR;
* Subjects with a history of primary or recurrent FSGS, membranous glomerulonephritis (MGN) or membranoproliferative glomerulonephritis (MPGN);
* Evidence of any active systemic or localized major infection;
* Use of any investigational drug or treatment up to 4 weeks before enrollment;
* Immunosuppressive therapies other than those described by this protocol;
* Planned systemic treatment with voriconazole, cisapride or ketoconazole that will not be discontinued before randomization;
* Prior treatment with aminoglycosides, amphotericin B, cisplatin or other drugs associated with renal dysfunction that is not discontinued before screening;
* Subjects with a screening total white blood cell count (WBC) ≤ 2000/mm3, hemoglobin ≤ 10g/dL and platelet count ≤ 100000/mm3;
* TGO/AST, TGP/ALT and bilirubins with values three times higher than reference values;
* Fasting triglycerides ≥ 400 mg/dL, fasting total cholesterol ≥ 350 mg/dL or LDL-cholesterol ≥ 160mg/dL despite the use of optimal lipid-lowering therapy;
* History of malignancy within 3 years before enrollment other than adequately treated basal cell or squamous cell carcinoma of the skin;
* Subjects who are known to be human immunodeficiency virus (HIV) positive or hepatitis B positive;
* Chronic hepatic failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in viral load of hepatitis C virus at 12 months after randomization. | Baseline,Months 3, 6, 9 and 12 after randomization
  HCV viremia will be measured by polymerase chain reaction (PCR)

SECONDARY OUTCOMES:
Incidence of acute allograft rejection | Weeks 1, 2, 3, months 1, 3, 6, 9 and 12 after randomization
  All patients will perform at least 07 protocol visits and should be performed renal biopsy during screening phase and during the follow up if present renal dysfunction or proteinuria.
Incidence of significant infections | Weeks1, 2, 3 and months 1, 3, 6,9 and 12 after randomization
  During the study visits the patient will be evaluated by a doctor and it will perform blood tests to assess their clinical conditions.
Development of proteinuria | Months 1, 3, 6, 9 and 12 after randomization
  Spot urine sample for protein and creatinine will be performed.
Development of malignance | Weeks 1, 2, 3 and months 1, 3, 6, 9 and 12 after randomization
  Medical evaluation will be performed during the protocol visits and if necessary biopsy and exams of imaging to confirm any suspected.
Development of dyslipidemia | Months 1, 3, 6, 9 and 12 after randomization
  Lipid levels: total cholesterol, HLD, LDL and triglycerides will be performed.
Development of liver impairment | Months 1, 3, 6, 9, and 12 after randomization
  Blood chemistry: TGO/AST, TGP/ALT , GGT and alkaline phosphatase will be performed.
Development of post-transplant diabetes | Months 1, 3, 6, 9 and 12
  Blood chemistry: Glucose will be performed.
Development of hypertension | Weeks 1, 2, 3 and months 1, 3, 6, 9 and 12 after randomization
  Vital signs will be performed
Graft loss survival | Weeks 1, 2 , 3 and months 1, 3 ,6, 9 and 12 after randomization
  Graft survival will be evaluated by our team doctor.
Patient survival | Weeks 1, 2, 3 and months 1, 3, 6, 9 and 12 after randomization
  Subject survival will be evaluated by our team doctor

CONTACTS AND LOCATIONS:
Overall Officials: Valter Garcia, Physician, Principal Investigator — IRMANDADE DA SANTA CASA DE MISERICÓRDIA DE PORTO ALEGRE; ELIZETE KEITEL, Physician, Study Chair — IRMANDADE DA SANTA CASA DE MISERICÓRDIA DE PORTO ALEGRE; MARIANA F RODRIGUES, PHARMACIST, Study Director — IRMANDADE DA SANTA CASA DE MISERICÓRDIA DE PORTO ALEGRE; DIEGO GNATTA, PHARMACIST, Study Director — IRMANDADE DA SANTA CASA DE MISERICÓRDIA DE PORTO ALEGRE; LARISSA S PACHECO, PHARMACIST, Study Director — IRMANDADE DA SANTA CASA DE MISERICÓRDIA DE PORTO ALEGRE; BRUNA D CARDOSO, PHARMACIST, Study Director — IRMANDADE DA SANTA CASA DE MISERICÓRDIA DE PORTO ALEGRE; RONIVAN L DAL PRA, PHARMACIST, Study Director — IRMANDADE DA SANTA CASA DE MISERICÓRDIA DE PORTO ALEGRE
Locations (1):
- Irmandade Da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Benedetto, F. D.; Sandro, S. D.; Ballarin, R.; Guaraldi, G.; Gerunda, G. E. Rapamycin and HIV Replication in Liver Transplant Recipients. Transplantation, 9, 1040, 2010.
- [Background] Boletis JN, Iniotaki-Theodoraki A, Psichogiou M, Stamatiadis DN, Viglis JV, Kostakis A, Stavropoulos-Giokas C. Immune status in renal transplant recipients with hepatitis C virus infection. Transplant Proc. 2002 Dec;34(8):3205-8. doi: 10.1016/s0041-1345(02)03656-4. No abstract available. PMID 12493421
- [Background] Gallego R, Henriquez F, Oliva E, Camacho R, Hernandez R, Hortal L, Sablon N, Quintana B, Santana R, Gonzalez F, Palop L, Vega N. Switching to sirolimus in renal transplant recipients with hepatitis C virus: a safe option. Transplant Proc. 2009 Jul-Aug;41(6):2334-6. doi: 10.1016/j.transproceed.2009.06.064. PMID 19715912
- [Background] Ingsathit A, Thakkinstian A, Kantachuvesiri S, Sumethkul V. Different impacts of hepatitis B virus and hepatitis C virus on the outcome of kidney transplantation. Transplant Proc. 2007 Jun;39(5):1424-8. doi: 10.1016/j.transproceed.2007.02.068. PMID 17580153
- [Background] Mas V, Alvarellos T, Chiurchiu C, Camps D, Massari P, de Boccardo G. Hepatitis C virus infection after renal transplantation: viral load and outcome. Transplant Proc. 2001 Feb-Mar;33(1-2):1791-3. doi: 10.1016/s0041-1345(00)02682-8. No abstract available. PMID 11267514
- [Background] Meier-Kriesche HU, Ojo AO, Hanson JA, Kaplan B. Hepatitis C antibody status and outcomes in renal transplant recipients. Transplantation. 2001 Jul 27;72(2):241-4. doi: 10.1097/00007890-200107270-00013. PMID 11477346
- [Background] Wagner D, Kniepeiss D, Schaffellner S, Jakoby E, Mueller H, Fahrleitner-Pammer A, Stiegler P, Tscheliessnigg KH, Iberer F. Sirolimus has a potential to influent viral recurrence in HCV positive liver transplant candidates. Int Immunopharmacol. 2010 Aug;10(8):990-3. doi: 10.1016/j.intimp.2010.05.006. Epub 2010 May 17. PMID 20483386